CLINICAL TRIAL: NCT03819803
Title: Fecal Microbiota Transplantation in Patients With Acute Gastrointestinal Graft-versus-host-disease After Allogeneic Stem Cell Transplantation
Brief Title: Fecal Microbiota Transplantation in aGvHD After ASCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI-aGvHD_01
Record Dates: First submitted 2018-09-14; First posted 2019-01-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Graft Versus Host Disease in GI Tract
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Patients with acute gastrointestinal graft-versus-host disease refractory to steroid treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Steroid refractory GI-aGvHD (Experimental): Patients with GI-aGvHD not sufficiently responding to GvHD therapy with corticosteroids.
  Intervention: Fecal microbiota transplantation
  Interventions: Biological: Fecal microbiota transplantation

INTERVENTIONS:
Biological: Fecal microbiota transplantation — 200 ml of a tested stool suspension of a healthy donor is instilled into the patient´s caecum or terminal ileum

SUMMARY:
Acute graft-versus-host-disease (aGvHD) is a typical complication after allogeneic hematopoetic stem cell transplantation (ASCT). About 30-60% of patients after ASCT are affected by aGvHD, which constitutes a relevant burden of morbidity and mortality in these patients.

Fecal microbiota transplantation (FMT) is a therapeutic concept to treat intestinal dysbiosis of various origin by infusion of the stool microbiota of a healthy donor into the gastrointestinal tract (GI) of a patient. FMT can be performed endoscopically by colonoscopic deployment of the donor microbiota into the patient´s caecum and terminal ileum.

Patients with gastrointestinal aGvHD (GI-aGvHD) are known to comprise a significant dysbiotic colonic microbiota that can be attenuated by FMT.

ELIGIBILITY:
Inclusion Criteria:

* first episode of histologically confirmed, steroid-refractory GI-aGvHD
* reduced bacterial diversity in the patient´s stool microbiota evidenced by 16s-rDNA measurement
* eligibility for repeated colonoscopic procedures
* informed consent

Exclusion Criteria:

* complications during a previous colonoscopy
* recurrent episode of GI-aGvHD
* lacking cardiopulmonary fitness for repeated colonoscopic procedures
* septic infection
* acute extraintestinal organ failure (excluding bone marrow)
* mechanical ileus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
GI-aGvHD remission | 90 days after first FMT
  Sustained remission of GI-aGvHD (CR or PR)

SECONDARY OUTCOMES:
GI-aGvHD remission | 45, 180 and 365 days after first FMT
  Sustained remission of GI-aGvHD (CR or PR)
Disease-free survival | 180 and 365 days after first FMT
  GI-aGvHD free survival
Recurrence of GI-GvHD | 365 days after remission
  Recurrence of GI-GvHD
Patient survival | 180 and 365 days after first FMT
  Survival (death or alive)
SUSAR (Suspected Unexpected Serious Adverse Reaction) | within 48 hours after a FMT
  Number of lethal or non-lethal SUSAR's
SAE (Serious Adverse Event) | within 48 hours after a FMT
  Number of lethal or non-lethal SAE's

CONTACTS AND LOCATIONS:
Overall Officials: Peter Prof. Dr. Neumeister, Principal Investigator — Department of Internal Medicine, Division of Hematology, Medical University of Graz
Locations (1):
- Division of Gastroenterology and Hepatology, Department of Internal Medicine, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No